CLINICAL TRIAL: NCT02581033
Title: Determinants of Sustained Virological Response After Discontinuation of Long-term Nucleoside Analogue Therapy in Chronic Hepatitis B Patients
Brief Title: Determinants of Virological Response After Discontinuation of Nucleoside Analogue Therapy in Hepatitis B Patients
Acronym: STOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Vincent's Hospital Melbourne (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Alexander Thompson, Professor, St Vincent's Hospital Melbourne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 032/14 Protocol # :APP106653
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Hepatitis B.
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nucleoside analogue therapy cessation (Experimental): To determine if a sustained virological response can be achieved after discontinuation of long-term nucleoside analogue therapy in chronic hepatitis B patients.
  Interventions: Drug: Nucleoside Analogue therapy

INTERVENTIONS:
Drug: Nucleoside Analogue therapy — Determinants of sustained virological response after discontinuation of long-term nucleoside analogue therapy in chronic hepatitis B patients.
  Other Names: Cessation of Nucleoside Analogue Therapy

SUMMARY:
Evaluation of the rate of sustained virological response among HBeAg-negativechronic hepatitis B patients who discontinue long-term NA therapy.

During this study participants will cease their prescribed medications, this will occur with immediate effect once enrolled into the study. The duration of cessation will be indefinite, unless clinically indicated for NA therapy re-start. Participants will be monitored as per protocol following cessation, monitoring will be by clinic visit and through blood test to monitor virological response. Clinical visits will be at the intervals of week 2, week, 4, week 8, week 12, week 18, following this they will be every 3 months out to 2 years when the participant will have completed the trial. Once the participant has completed the trial they will not commence again, the aim is for an indefinite cessation of NA therapy.

DETAILED DESCRIPTION:
During this study participants will cease their prescribed medications, this will occur with immediate effect once enrolled into the study. The duration of cessation will be indefinite, unless clinically indicated for NA therapy re-start. Participants will be monitored as per protocol following cessation, monitoring will be by clinic visit and through blood test to monitor virological response. Clinical visits will be at the intervals of week 2, week, 4, week 8, week 12, week 18, following this they will be every 3 months out to 2 years when the participant will have completed the trial. Once the participant has completed the trial they will not commence again, the aim is for an indefinite cessation of NA therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, age >18 years
* Subjects must be able to understand and agree to comply with the prescribed intervention (NA cessation), visits and reliably communicate with study personal about adverse events
* Able to provide informed consent.
* Chronic Hepatitis B virus infection
* HBeAg negative at time if initiation of NA therapy
* Meet current APASL guidelines for consideration of antiviral cessation:
* uninterrupted NA treatment for >2 years and
* undetectable serum HBV DNA on three separate occasions >= 6 months apart (undetectable defined by a value < lower limit of detection using a sensitive commercial PCR assay)
* Normal serum ALT levels (according to the uppers limit of normal of the local laboratory)
* Minimal to moderate liver fibrosis defined as:
* METAVIR liver fibrosis stage F0-F3 inclusive prior to initial NA therapy and/or
* Transient liver elastogram (TLE) (Fibroscan) < /= 9.6 kPa at screening

Exclusion Criteria:

* HBeAg positive chronic hepatitis B at the time of NA initiation
* HBV associated extra hepatic manifestations
* Documented or suspected hepatocellular carcinoma (HCC)
* History of decompensated liver disease
* Compensated cirrhosis defined as:
* METAVIR liver fibrosis stage 4 on pre-treatment biopsy; OR
* TLE > 9.6 kPa at screening
* Co-infection with HIV,HCV or HDV
* Latrogenic or disease related immunosuppression (e.g. treatment with systemic glucocorticoids, TNFa-antibodies, and other immunosuppressive drugs)
* Significant alcohol consumption (> 30 g/day for women and > 50 g/day for men)
* Current known history of cancer within 5 years of screening
* Pregnant or breast feeding
* Other known significant liver disease (including but not limited to haemochromatosis, autoimmune hepatitis, alcoholic liver disease)
* Participation in any other interventional trial
* Poor Venous access
* Suspected lack of compliance
* Any medical or social reason which in the opinion of the investigator would make the subject inappropriate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The primary aim of this study is to evaluate the rate of sustained virological response among HBeAg-negative chronic hepatitis B patients who discontinue long-term NA therapy. The outcome is to be assessed by serum assay. | Patients will be closely followed for 2 years prospectively, at the following time points; 2 weeks post cessation, 4 weeks, 8 weeks, 12 weeks, 18 weeks, then from 6 months the visits will be 3 monthly out to two years, to observe for virological changes.

SECONDARY OUTCOMES:
To identify novel immunological determinants of SVR, the assessment will be by serum assay. | Patients will be closely followed for 2 years prospectively, at the following time points; 2 weeks post cessation, 4 weeks, 8 weeks, 12 weeks, 18 weeks, then from 6 months the visits will be 3 monthly out to two years.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Thompson, MD, Principal Investigator — St Vincent's Hospital Melbourne
Locations (1):
- St Vincent's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hume SJ, Hall S, Burns G, Vogrin S, Tassone D, Desmond P, Ratnam D, Levy MT, Sawhney R, Nicoll A, Valaydon Z, Strasser SI, Ngu M, Sinclair M, Meredith C, Matthews GV, Visvanathan K, Holmes JA, Thompson AJ. Long-Term Follow-Up of Patients in a Prospective Study of NA Discontinuation Identifies Different Patterns of HBsAg Loss. Aliment Pharmacol Ther. 2026 Jan;63(2):231-241. doi: 10.1111/apt.70332. Epub 2025 Aug 21. PMID 40842267